CLINICAL TRIAL: NCT01295515
Title: Effect of Interferon Alpha 2b Intensification on HIV-1 Residual Viremia in Individuals Suppressed on Antiretroviral Therapy
Brief Title: Interferon Alpha 2b Intensification in HIV-Positive Individuals on Antiretroviral Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Frank Maldarelli, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110057; 11-I-0057 (Other: NIH)
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: HIV Infection
Keywords: HIV; Replication; Antiretroviral; Interferon; Reservoirs
MeSH Terms: conditions — HIV Infections | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Interferon treatment (Experimental): Interferon treatment The intervention is administration of Pegylated Interferon Alpha 2b (PEGINTRON) weekly for four weeks
  Interventions: Drug: Pegylated Interferon Alpha 2b (PEGINTRON)

INTERVENTIONS:
Drug: Pegylated Interferon Alpha 2b (PEGINTRON) — pegylated preparation of interferon alpha 2b
  Other Names: PEGINTRON

SUMMARY:
Background:

* Antiretroviral therapy (ART) has been able to improve the lifespan of individuals infected with human immunodeficiency virus type 1 (HIV-1), but ART requires continuous treatment that has substantial consequences on quality of life. Recent research is attempting to determine whether this persistent infection stems from a low-level infection where new cells are continually infected with HIV, or from cells that live for a long time after infection. ART is very active against the virus in new cells, but has no effect on long-lived cells that are already infected with HIV-1 at the start of ART. As a result, new strategies may be necessary to reduce or eradicate these 'reservoir' cells.
* Interferon is a natural substance made by the body to combat virus infections, and can be made as an injectable drug known as PEGINTRON. Researchers are interested in determining whether PEGINTRON therapy will also reduce the residual low levels of HIV in patients who are already taking ART.

Objectives:

- To evaluate the effectiveness of PEGINTRON injections on HIV levels in participants currently undergoing antiretroviral therapy.

Eligibility:

- Individuals at least 18 years of age who have been diagnosed with HIV, are currently undergoing antiretroviral therapy, and have maintained HIV virus blood counts that are not detectable by current commercial tests for at least 12 months before the start of the study.

Design:

* This study will involve separate screening and treatment processes.
* Participants will be screened with a physical examination and medical history, including blood and urine samples. The screening analysis to determine study eligibility will take several weeks. Participants will have apheresis to provide sufficient numbers of blood cells for evaluation by the study researchers.
* Eligible participants will begin a 4-week course of PEGINTRON injections using the standard dose of PEGINTRON that is approved for treatment of chronic hepatitis C. Participants will have weekly injections and have frequent blood tests to measure HIV virus levels.
* Participants who experience problems in maintaining safe numbers of white blood cells during the study may receive injections of filgrastim to increase their white blood cell count.
* After the 4 weeks of treatment, participants will return for additional blood tests on study days 28, 35, 42, 49, 56, and 84, and Weeks 16, 24, 36, and 48 (i.e., through the end of 1 year after the start of the study).

DETAILED DESCRIPTION:
As a result of combination antiretroviral therapy (ART), morbidity and mortality from acquired immunodeficiency syndrome has declined significantly in the past 15 years, at least in developed countries. Human immunodeficiency virus type 1 (HIV-1) infected individuals now live longer, but must undergo continuous therapy that has substantial consequences on quality of life.

ART suppresses HIV-1 viremia below the limits of detection in current commercial assays (c. 50 copies/mL plasma), but HIV viremia persists even after prolonged suppressive therapy. The origin of this residual viremia is yet not clear, but data suggest that production from long lived HIV infected cells may contribute to viremia.

Antiretrovirals are extremely active against replicating cells, and can thus successfully stop viral replication, but have no effect on long-lived viral reservoirs of cells already infected with HIV-1 at the time antiretroviral therapy is initiated. As a result, new strategies are necessary to reduce or eradicate long-lived reservoirs.

Interferon alpha is a natural cytokine with antiviral activity. Prior to the introduction of antiretroviral therapy, several studies demonstrated modest effect of interferon alpha in HIV-1 viremia in active cycles of infection in infected individuals. Interferon alpha was also effective in vitro in decreasing virus production from cells chronically infected with HIV-1. With the introduction of potent antiretroviral therapy, interferon was not developed as a direct anti-HIV drug. Interferon alpha is relatively effective in therapy of hepatitis C virus (HCV) infection, and has been used in HIV-1/HCV coinfected individuals. Kottilil and coworkers in the Laboratory of Immunoregulation National Institute of Allergy and Infectious Diseases (NIAID) have shown a decrease in HIV-1 ribonucleic acid (RNA) levels in HCV coinfected participants treated with pegylated interferon alpha and ribavirin. In stored samples from that study, we conducted a retrospective trial on samples from participants with HIV-1 RNA levels of <50 copies/mL, showing a further reduction in residual viremia using an ultrasensitive Single Copy Assay (SCA) developed in our laboratory. As such the effects of interferon on HIV viremia and cell associated HIV RNA are of growing interest.

In this protocol we will conduct a prospective, non-randomized, single arm, pilot study to investigate the effect of pegylated interferon alpha 2b on HIV-1 RNA levels as an additional drug in participants undergoing suppressive antiretroviral therapy with viral RNA levels suppressed to less than 50 copies/mL plasma. As patients may have levels of HIV RNA that are lower than our limit of detection, we will also investigate levels of HIV nucleic acid species in cells as well. We will determine whether interferon alpha therapy will reduce residual viremia or cell associated HIV RNA in participants on suppressive ART, which will expand our understanding of persistent low-level viremia and the pathogenesis of HIV in infected individuals.

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible for study participation, a volunteer must satisfy all of the following inclusion criteria:

1. Age greater than or equal to 18 years.
2. Documentation of human immunodeficiency virus type 1 (HIV-1) infection by any licensed enzyme-linked immunosorbent assay (ELISA) test and confirmed by a Western Blot.
3. Receiving a Department of Health and Human Services (DHHS)-approved antiretroviral (ARV) regimen.
4. Level of cell-associated HIV ribonucleic acid (RNA) greater than or equal to 5 copies/million peripheral blood mononuclear cells (PBMC) done at screening visit 1.
5. HIV-1 RNA levels less than detectable by current commercial means (e.g., Roche Amplicor, b-deoxyribonycleic acid (DNA) test) for a minimum of 12 months prior to screening at all time points, and with at least 2 measurements in this 12 month window.
6. Cluster of differentiation 4 (CD4) greater than or equal to 300 cells/mm(3) at pre-entry visit within 14 days prior to enrollment.
7. Ability to sign informed consent and willingness to comply with the study requirements and clinic policies.
8. No evidence of viral hepatitis co-infection as assessed by Hepatitis C antibody, HCV RNA, and hepatitis B surface antigen; determinations at pre-entry visit within 28 days prior to enrollment.
9. No history of or evidence of autoimmune hepatitis or other autoimmune disorders at screening, or Antinuclear antibody (ANA > 3 times upper limit of normal.
10. Laboratory values at pre-entry visit within 14 days prior to enrollment:

    * Alkaline phosphatase <2.0 times upper limit of normal
    * Alanine transaminase (ALT) <2.0 times upper limit of normal
    * Total bilirubin < 2.5 mg/dL (< 40 mg/dL if on Atazanavir)
    * Creatinine clearance greater than or equal to 60 mL/min as estimated by the Cockcroft-Gault equation
    * Neutrophil count greater than or equal 1500 cells/mm(3)
    * Platelets greater than or equal to 150,000/ mm(3)
    * Hemoglobin greater than or equal to 12.0 mg/dL for men and >11.0 g/dL for women
    * Fasting glucose < 126 mg/dL
11. No history or evidence of significant clinical depression at screening that in the opinion of the investigator would affect the ability of the patient to participate in the study, or which would constitute a threat for his/her health in case of relapse upon interferon (INF) treatment. The Beck Depression Inventory score must be less than or equal to 13 at pre-entry visit.
12. No history of INF/pegylated interferon (PEG-INF) therapy.
13. If capable of pregnancy: use of effective contraception during study: effective contraception methods include abstinence, surgical sterilization of either partner, barrier methods such as diaphragm, condom, cap or sponge, or use of hormonal contraception with an anti-HIV regimen that will not alter metabolism of hormonal contraception.
14. Participants must have primary medical care outside this protocol: participants will have to provide Primary Care Doctors contact information.

EXCLUSION CRITERIA:

A volunteer will be ineligible to participate in this study if any of the following criteria are met:

1. History of neoplastic disease requiring cytotoxic therapy including hydroxyurea.
2. Use of long-term systemic corticosteroids, immunosuppressive agents, or cytotoxic agents within 60 days prior to enrollment.
3. Any vaccination within 30 days prior to enrollment. Individuals interested in participating who require vaccination will delay screening until 30 day period is completed.
4. Concurrent therapy with investigational cytokines including interleukin-2 (IL-2) or interleukin-12 (IL-12) during the course of the study. Prior administration of cytokines is not an exclusion criterion; at least 4 months from most recent cycle of IL-2 or IL-12 is required.
5. Any febrile illness (>38 degrees C) in the 3 weeks prior to enrollment or any acute therapy for a serious infection completed within 30 days prior to enrollment.
6. Current pregnancy or lactation, history of pregnancy in the last 4 months.
7. Preexisting autoimmune disorders including inflammatory bowel diseases, psoriasis, idiopathic thrombocytopenic purpura, lupus erythematous, autoimmune hemolytic anemia, scleroderma, severe psoriasis, rheumatoid arthritis, and optic neuritis.
8. History of severe retinopathy or evidence of severe retinopathy judged by pre-entry ophthalmologic examination.
9. Known allergy/sensitivity to study drug or its formulation.
10. History of seizure disorders or current anticonvulsant use.
11. Any history of medical conditions associated with chronic liver disease (genetic hemochromatosis, alcoholic liver disease, toxin exposures, and autoimmune hepatitis) or documented cirrhosis due to any cause.
12. History of pulmonary disease associated with functional limitation.
13. Documented history of thyroid disease.
14. Active drug or alcohol use or dependence, which in the opinion of the investigator, would interfere with complying with the study requirements.
15. Known hypersensitivity to Escherichia coli-derived products such as filgrastim.
16. Any systemic illness that will make it unlikely that the subject will be able to return for the required study visits.
17. History of, or any condition that in the opinion of the investigator would interfere with the conduct of the study, or it would not be in the best interest of the subject to enroll in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2011-02-11 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Maldarelli, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palmer S, Maldarelli F, Wiegand A, Bernstein B, Hanna GJ, Brun SC, Kempf DJ, Mellors JW, Coffin JM, King MS. Low-level viremia persists for at least 7 years in patients on suppressive antiretroviral therapy. Proc Natl Acad Sci U S A. 2008 Mar 11;105(10):3879-84. doi: 10.1073/pnas.0800050105. Epub 2008 Mar 10. PMID 18332425
- [Background] Maldarelli F, Palmer S, King MS, Wiegand A, Polis MA, Mican J, Kovacs JA, Davey RT, Rock-Kress D, Dewar R, Liu S, Metcalf JA, Rehm C, Brun SC, Hanna GJ, Kempf DJ, Coffin JM, Mellors JW. ART suppresses plasma HIV-1 RNA to a stable set point predicted by pretherapy viremia. PLoS Pathog. 2007 Apr;3(4):e46. doi: 10.1371/journal.ppat.0030046. PMID 17411338
- [Background] Dinoso JB, Kim SY, Wiegand AM, Palmer SE, Gange SJ, Cranmer L, O'Shea A, Callender M, Spivak A, Brennan T, Kearney MF, Proschan MA, Mican JM, Rehm CA, Coffin JM, Mellors JW, Siliciano RF, Maldarelli F. Treatment intensification does not reduce residual HIV-1 viremia in patients on highly active antiretroviral therapy. Proc Natl Acad Sci U S A. 2009 Jun 9;106(23):9403-8. doi: 10.1073/pnas.0903107106. Epub 2009 May 22. PMID 19470482
- [Result] Somsouk M, Dunham RM, Cohen M, Albright R, Abdel-Mohsen M, Liegler T, Lifson J, Piatak M, Gorelick R, Huang Y, Wu Y, Hsue PY, Martin JN, Deeks SG, McCune JM, Hunt PW. The immunologic effects of mesalamine in treated HIV-infected individuals with incomplete CD4+ T cell recovery: a randomized crossover trial. PLoS One. 2014 Dec 29;9(12):e116306. doi: 10.1371/journal.pone.0116306. eCollection 2014. PMID 25545673
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-I-0057.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Interferon Treatment: Interferon treatment
  Pegylated Interferon Alpha 2b (PEGINTRON): pegylated preparation of interferon alpha 2b
Period: Overall Study
Arm/Group | Interferon Treatment
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: HIV-infected individuals undergoing antiretroviral therapy
Arm/Group | Interferon Treatment
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.85 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 5
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Pre- and Post- Interferon Alpha on Human Immunodeficiency Virus Type 1 (HIV-1) Ribonucleic Acid (RNA)
Description: Cell associated HIV nucleic acid levels were measured using a single copy assay, and numbers of cells were quantified using a polymerase chain reaction method that detects RNA.
Time Frame: week 4 (post) compared to week 0 (pre)
Population: A total of 7 participants were analyzed overall and each row of data represents each participant's analyzed data.
Measure: Number; unit: # of copies of HIV RNA/million cells
Arm/Group | Interferon Treatment
Number analyzed (Participants) | 7
# of copies of HIV RNA/million cells
  Patient #1 HIV RNA Pre: number analyzed (Participants) | 1
  Patient #1 HIV RNA Pre | 670
  Patient #1 HIV RNA Post: number analyzed (Participants) | 1
  Patient #1 HIV RNA Post | 180
  Patient #2 HIV RNA Pre: number analyzed (Participants) | 1
  Patient #2 HIV RNA Pre | 90
  Patient #2 HIV RNA Post: number analyzed (Participants) | 1
  Patient #2 HIV RNA Post | 130
  Patient #3 HIV RNA Pre: number analyzed (Participants) | 1
  Patient #3 HIV RNA Pre | 810
  Patient #3 HIV RNA Post: number analyzed (Participants) | 1
  Patient #3 HIV RNA Post | 420
  Patient #4 HIV RNA Pre: number analyzed (Participants) | 1
  Patient #4 HIV RNA Pre | 450
  Patient #4 HIV RNA Post: number analyzed (Participants) | 1
  Patient #4 HIV RNA Post | 390
  Patient #5 HIV RNA Pre: number analyzed (Participants) | 1
  Patient #5 HIV RNA Pre | 12
  Patient #5 HIV RNA Post: number analyzed (Participants) | 1
  Patient #5 HIV RNA Post | 51
  Patient #6 HIV RNA Pre: number analyzed (Participants) | 1
  Patient #6 HIV RNA Pre | 850
  Patient #6 HIV RNA Post: number analyzed (Participants) | 1
  Patient #6 HIV RNA Post | 300
  Patient #7 HIV RNA Pre: number analyzed (Participants) | 1
  Patient #7 HIV RNA Pre | 250
  Patient #7 HIV RNA Post: number analyzed (Participants) | 1
  Patient #7 HIV RNA Post | 310

2. Secondary Outcome: Fold Change in Ribonucleic Acid (RNA) and Deoxyribonucleic Acid (DNA) in Human Immunodeficiency Virus Type 1 (HIV-1) Genetic Variation in Individuals Undergoing Interferon Therapy
Description: The outcome measure is the fold change in the ratio of HIV RNA to HIV DNA. For the pre and post interferon time point, the level of HIV RNA is divided by the level of HIV DNA and this ratio of the HIV RNA/DNA pre and post interferon is calculated to yield the fold change in HIV RNA/DNA levels. Fold change does not have units.
Time Frame: week 4 (post) and week 0 (pre)
Population: A total of 7 participants were analyzed overall and each row of data represents each participant's analyzed data.
Measure: Number; unit: fold change
Arm/Group | Interferon Treatment
Number analyzed (Participants) | 7
fold change
  Patient #1: number analyzed (Participants) | 1
  Patient #1 | 0.408
  Patient #2: number analyzed (Participants) | 1
  Patient #2 | 1.44
  Patient #3: number analyzed (Participants) | 1
  Patient #3 | 0.684
  Patient #4: number analyzed (Participants) | 1
  Patient #4 | 1.12
  Patient #5: number analyzed (Participants) | 1
  Patient #5 | 2.24
  Patient #6: number analyzed (Participants) | 1
  Patient #6 | 4.37
  Patient #7: number analyzed (Participants) | 1
  Patient #7 | 1.05

3. Secondary Outcome: Pre-and Post- Plasma Human Immunodeficiency Virus (HIV) Ribonucleic Acid (RNA) in HIV-infected Individuals
Description: The outcome measure is copies of HIV RNA per ml of plasma. HIV RNA levels are measured using a polymerase chain reaction method.
Time Frame: week 4 (post) compared to week 0 (pre)
Population: Median and standard deviation were calculated using multiple samples from each participant. On patient #5 there was an error with the machine when the samples were ran and they did not have any other samples to rerun it. Patient #5 will not be analyzed since there is no more samples.
Measure: Median (Standard Deviation); unit: copies/ml
Arm/Group | Interferon Treatment
Number analyzed (Participants) | 6
copies/ml
  Patient #1 Pre: number analyzed (Participants) | 1
  Patient #1 Pre | 0.7 (0.8)
  Patient #1 Post: number analyzed (Participants) | 1
  Patient #1 Post | 3.8 (1.9)
  Patient #2 Pre: number analyzed (Participants) | 1
  Patient #2 Pre | 0.2 (0.4)
  Patient #2 Post: number analyzed (Participants) | 1
  Patient #2 Post | .02 (0)
  Patient #3 Pre: number analyzed (Participants) | 1
  Patient #3 Pre | 3.8 (1.9)
  Patient #3 Post: number analyzed (Participants) | 1
  Patient #3 Post | 0.8 (0.9)
  Patient #4 Pre: number analyzed (Participants) | 1
  Patient #4 Pre | .02 (0)
  Patient #4 Post: number analyzed (Participants) | 1
  Patient #4 Post | 1.5 (1.2)
  Patient #6 Pre: number analyzed (Participants) | 1
  Patient #6 Pre | 1.3 (1.1)
  Patient #6 Post: number analyzed (Participants) | 1
  Patient #6 Post | 0.36 (0.6)
  Patient #7 Pre: number analyzed (Participants) | 1
  Patient #7 Pre | 9.1 (3.0)
  Patient #7 Post: number analyzed (Participants) | 1
  Patient #7 Post | 8.8 (3.0)

4. Secondary Outcome: Count of Participants With Serious and Non-serious Adverse Events Assessed by the Division of Acquired Immune Deficiency Syndrome (AIDS) Table for Grading Adult Adverse Events.
Description: Here is the count of participants with serious and non-serious adverse events assessed by the Division of Acquired Immune Deficiency Syndrome (AIDS) Table for Grading Adult Adverse Events for severity (mild/moderate/severe), expectedness (expected/unexpected), and relatedness to study drug (definitely, probably, possibly, unlikely, or unrelated).
Time Frame: Date consent signed to date off study, approximately 66 months and 2 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Interferon Treatment
Number analyzed (Participants) | 7
Participants | 7

5. Primary Outcome: Pre- and Post- Interferon Alpha on Human Immunodeficiency Virus Type 1 (HIV-1) Deoxyribonucleic Acid (DNA)
Description: Cell associated HIV nucleic acid levels were measured using a single copy assay, and numbers of cells were quantified using a polymerase chain reaction method that detects C-C chemokine receptor type 5 (CCR5) DNA.
Time Frame: week 4 (post) compared to week 0 (pre)
Population: A total of 7 participants were analyzed overall and each row of data represents each participant's analyzed data.
Measure: Number; unit: # of copies of DNA/million cells
Arm/Group | Interferon Treatment
Number analyzed (Participants) | 7
# of copies of DNA/million cells
  Patient #1 HIV DNA Pre: number analyzed (Participants) | 1
  Patient #1 HIV DNA Pre | 1200
  Patient #1 HIV DNA Post: number analyzed (Participants) | 1
  Patient #1 HIV DNA Post | 790
  Patient #2 HIV DNA Pre: number analyzed (Participants) | 1
  Patient #2 HIV DNA Pre | 150
  Patient #2 HIV DNA Post: number analyzed (Participants) | 1
  Patient #2 HIV DNA Post | 150
  Patient #3 HIV DNA Pre: number analyzed (Participants) | 1
  Patient #3 HIV DNA Pre | 660
  Patient #3 HIV DNA Post: number analyzed (Participants) | 1
  Patient #3 HIV DNA Post | 500
  Patient #4 HIV DNA Pre: number analyzed (Participants) | 1
  Patient #4 HIV DNA Pre | 400
  Patient #4 HIV DNA Post: number analyzed (Participants) | 1
  Patient #4 HIV DNA Post | 310
  Patient #5 HIV DNA Pre: number analyzed (Participants) | 1
  Patient #5 HIV DNA Pre | 10
  Patient #5 HIV DNA Post: number analyzed (Participants) | 1
  Patient #5 HIV DNA Post | 19
  Patient #6 HIV DNA Pre: number analyzed (Participants) | 1
  Patient #6 HIV DNA Pre | 520
  Patient #6 HIV DNA Post: number analyzed (Participants) | 1
  Patient #6 HIV DNA Post | 420
  Patient #7 HIV DNA Pre: number analyzed (Participants) | 1
  Patient #7 HIV DNA Pre | 390
  Patient #7 HIV DNA Post: number analyzed (Participants) | 1
  Patient #7 HIV DNA Post | 460

ADVERSE EVENTS:
Time Frame: The adverse events were collected from date of consent to date off study, approximately 66 months and 2 days.
Description: Adverse events were graded according to the Division of Acquired Immune Deficiency Syndrome (AIDS) Table for Grading Adults Adverse Events.
Arm/Group | Interferon Treatment
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon Treatment (N=7)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon Treatment (N=7)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Alanine aminotransferase increased (Investigations) | 2 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (7)
Aspartate aminotransferase increased (Investigations) | 2 (4)
Blood cholesterol increased (Investigations) | 1 (1)
Blood pressure increased (Vascular disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Dermatophytosis (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (3)
Dry mouth (Gastrointestinal disorders) | 2 (4)
Fatigue (General disorders) | 3 (7)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Hemoglobin decreased (Investigations) | 1 (1)
Headache (Nervous system disorders) | 2 (7)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Injection site erythema (Injury, poisoning and procedural complications) | 1 (1)
Injection site reaction (Injury, poisoning and procedural complications) | 2 (3)
Injury (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (12)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Neutrophil count decreased (Investigations) | 5 (10)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Platelet count decreased (Investigations) | 2 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Prothrombin time prolonged (Investigations) | 1 (1)
Pyrexia (General disorders) | 4 (6)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
White blood cell count decreased (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form: Screening consent (2015-05-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT01295515/ICF_000.pdf
  • Informed Consent Form: Standard consent (2015-05-18): https://cdn.clinicaltrials.gov/large-docs/15/NCT01295515/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2015-03-31): https://cdn.clinicaltrials.gov/large-docs/15/NCT01295515/Prot_SAP_002.pdf